CLINICAL TRIAL: NCT05320809
Title: A Phase I Study to Evaluate the Safety and Immunogenicity of 3D189 in Patients With Hematologic Malignancies
Brief Title: Study of 3D189 in Patients With Hematologic Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 3D Medicines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3D189-CN-001
Record Dates: First submitted 2022-03-19; First posted 2022-04-11 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-11

CONDITIONS: Acute Leukemia; Multiple Myeloma; Non-Hodgkin Lymphoma; Higher-risk Myelodysplastic Syndrome
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 3D189 (Experimental)
  Interventions: Biological: 3D189

INTERVENTIONS:
Biological: 3D189 — 3D189 (200 mcg per peptide x 4 WT1 peptides within the drug product; total weight: 800 mcg) is mixed (1:1 v/v) and emulsified with the adjuvant Montanide, which is then injected subcutaneously to the patient.
  A maximum of 15 total injections of 3D189 will be administered as follows:
  1. Initial immunization induction phase（the first series of 6 injections of 3D189): every 2 weeks (Weeks 0 - 10) followed by a 4-week period of no treatment.
  2. Early immune booster phase（the second series of 6 injections of 3D189): every 4 weeks (between Weeks 14 and 34) followed by a 6-week period of no treatment.
  3. Late immune booster phase（the third series of 3 injections of 3D189): every 6 weeks (between Weeks 40 and 52).

SUMMARY:
To assess the safety, immunogenicity and preliminary efficacy of 3D189 in patients with hematological malignancies.

DETAILED DESCRIPTION:
This is a phase 1, open-label, non-comparative, multicenter study of 3D189 (also known as galinpepimut-S), a multivalent peptide vaccine targeting Wilms Tumor-1 (WT1), for maintenance immunotherapy in patients with WT1-positive hematological malignancies, including patients with acute leukemia (AL) patients in complete remission (CR), or multiple myeloma (MM), non-Hodgkin lymphoma (NHL) or higher-risk myelodysplastic syndrome (MDS) patients who have received at least first-line standard therapy and recently achieved CR or partial remission (PR), if the latter is the best achievable response for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to understand and provide signed informed consent for the study.
* Male or female patients ≥ 18 years of age on the day of signing informed consent.
* Have a histologically or cytologically confirmed hematological malignancy and have achieved complete remission (CR) or partial remission (PR) after at least one line of standard therapy, and are not suitable for hematopoietic stem cell transplant (HSCT) for the following reasons: a) not eligible for HSCT due to intercurrent medical conditions; b) lack of an available HLA-matched donor for allogeneic HSCT; c) not able to accept HSCT for financial reasons; d) without a potential indication for HSCT (e.g. having a relatively favorable prognosis or low risk of relapse). However, patients who have previously received autologous HSCT but remain MRD+ or in remission after salvage therapy for post-transplant relapse are allowed to be recruited.

Including the following 4 types of hematological malignancies:

1. Acute Leukemia (AL): including acute myeloma leukemia (AML) and acute lymphoblastic leukemia (ALL), in morphological complete remission with complete or incomplete blood count recovery (CR or CRi), and having completed any planned post-remission therapy;
2. Myelodysplastic Syndrome (MDS): Revised International Prognostic Scoring System (IPSS-R) risk score > 3.5, having achieved CR or PR following prior therapy;
3. Multiple Myeloma (MM): having achieved stringent complete response (sCR), CR or very good partial response (VGPR), or PR if deeper response cannot be obtained from adequate therapy.
4. Non-Hodgkin Lymphoma (NHL): preference for patients with diffuse large B-cell lymphoma (DLBCL) and follicular lymphoma (FL) who have achieved CR or PR following prior therapy.

   * Have a documented WT1 positive disease. This is defined as detectable presence of WT1 transcript via real-time quantitative polymerase chain reaction (RT-PCR) in patients'bone marrow or peripheral blood samples, or WT1 expression by immunohistochemistry (IHC) in archived (paraffin embedded, unstained slides) or freshly biopsied tumor tissues from bone marrow or lymph nodes or extranodal lesions ( for NHL patients).
   * Eastern Cooperative Oncology Group (ECOG) performance status of 0~1.
   * Estimated life expectancy ≥ 6 months.
   * The interval between the last antitumor therapy (including surgery, radiotherapy and systemic therapy) and the first study treatment must be at least 4 weeks or 10 half-lives of chemotherapy drugs (whichever is shorter), and the toxicity of the previous therapies have recovered to ≤ grade 1 [according to the Common Terminology Criteria for Adverse Events (CTCAE) 5.0], except for toxicity such as alopecia, which in the judgment of the investigator is not a safety risk.
   * Have adequate organ and bone marrow function, defined as follows:

1) Blood count (participants must not have received transfusion of blood products within 7 days prior to this test): hemoglobin (Hb) ≥ 9.0 g/dL; neutrophil (NEUT) ≥ 1.0×109/L; platelet (PLT) ≥ 50×109/L; 2) Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ×ULN (upper limit of normal); but for subjects with liver metastasis, ALT or AST ≤ 5×ULN; total bilirubin (TBIL) ≤ 1.5 × ULN, or TBIL > 1.5 × ULN, but direct bilirubin (DBIL) ≤ 1.0 × ULN; 3) Renal function: serum creatinine ≤ 1.5 × ULN or endogenous creatinine clearance rate ≥ 50 ml/min (Cockcroft-Gault formula); 4) Coagulation: international normalized ratio (INR) ≤ 1.5, activated partial thromboplastin time (APTT) ≤ 1.5 ×ULN, unless subjects are receiving anticoagulant therapy as long as INR or APTT is within the therapeutic range of intended use of anticoagulants; 5) Cardiac function: left ventricular ejection fraction (LVEF) ≥ 50% by echocardiography.

• Subjects (including partners) must agree to use an adequate method of contraception, starting with the screening visit through 4 months after the last dose of study treatment.

Exclusion Criteria:

* Previously treated with any therapy targeting WT1.
* Have known hypersensitivity to peptide biologics, or to immune adjuvants Montanide and/or GM-CSF.
* Subjects with acute promyelocytic leukemia (APL or M3).
* Presence of central nervous system (CNS) invasion and/or carcinomatous meningitis; participants with previously cured brain or meningeal metastasis can be allowed.
* Have undergone prior allogeneic HSCT, or plan to perform HSCT during the study period.
* Received live vaccine within 4 weeks prior to the first dose of study treatment.
* Currently participate in or have participated in a study of an interventional agent or device within 4 weeks prior to the first dose of study treatment.
* Have a known additional malignancies within the past 5 years, with the exception of cured skin basal cell carcinoma or cervical cancer in situ or other carcinoma in situ.
* Have an active autoimmune disease or any disease that requires long-term use of systemic corticosteroids (at doses greater than 10 mg daily of prednisone equivalent) or any other form of immunosuppressive agents, hormone replacement therapy for adrenocortical insufficiency, hypopituitarism, hypothyroidism, or type I diabetes mellitus is not considered a form of systemic treatment and is allowed.
* Have a diagnosis of primary immunodeficiency disease, or acquired immunodeficiency syndrome, or a positive test for human immunodeficiency virus (HIV).
* Presence of active tuberculosis.
* Have a history of a severe cardiovascular disease such as class III or IV heart failure [New York Heart Association (NYHA) criteria], myocardial infarction or stroke, unstable angina within 6 months prior to start of study treatment.
* QTcF interval tested during the screening period ≥ 450 msec (for male subjects) or ≥ 470 msec (for female).
* Have an acute severe infection requiring systemic therapy during the screening period.
* Positive for HBsAg and HBV DNA ≥ 103 IU/ml; or positive for HCV antibodies and HCV RNA level is above the detection limit.
* Are pregnant or breastfeeding, or have a positive serum pregnancy test during the screening period (for female subjects of childbearing potential).
* Have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Any condition, therapy or laboratory abnormality that, in the opinion of the investigator, might affect the participant's compliance, pose an unwarranted high risk to the participant, or interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number and frequency of TRAEs, including AE and SAEs (safety parameters) | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment, up to 13 months
  ncidence and severity of adverse events (AEs) and serious adverse events (SAEs) related to the study treatment (graded in accordance with National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0)
Immune response rate of 3D189 vaccination among subjects | From baseline (pre-treatment) to the end of study treatment,up to 12 months
  The rate of positive results for any of the immune tests used to assess the WT1 -specific T-cell immune responses.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 24 months
  From time of registration to the time of subject death.
Relapse-free survival (RFS) or progression-free survival (PFS) | up to 12 months
  From time of registration to the time of documented morphological leukemic relapse (for AL patients only) or disease progression (for MDS, MM and NHL patients) or subject death (for all patients)
Overall response rate (ORR) | up to 12 months
  Partial response (PR) or complete response (CR) in MDS, MM or NHL patients receiving 3D189 treatment, as evaluated by the investigators according to the corresponding response evaluation criteria and by comparison with baseline.
Duration of Response (DoR) | up to 12 months
  Time interval between the documentation of ORR (CR/PR) post study treatment and the documentation of progressive disease (PD) (for MDS, MM or NHL patients).
Disease control rate (DCR) | up to 12 months
  The percentage of patients who achieve CR or PR post study treatment or who remain stable for at least the first 12 weeks of study treatment (for MDS, MM or NHL patients).

CONTACTS AND LOCATIONS:
Overall Officials: jianxiang wang, Ph.D, Principal Investigator — Institute of Hematology & Blood Diseases Hospital,Chinese Academy of Medical Science & Peking Union Medical College
Locations (4):
- China (4):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical, Shengyang, Liaoning
  - Blood Disease Hospital , Chinese Academy of Medical Science, Tianjing, Tianjing

IPD SHARING:
Plan to Share IPD: No